CLINICAL TRIAL: NCT03501875
Title: Study of Coronary Calcification in Subjects With Autosomal Dominant Familial Hypercholesterolemia Heterozygous
Acronym: FH-CALC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institute of Cardiometabolism and Nutrition, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P170703J; 2017-A02904-49 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2018-03-02; First posted 2018-04-18 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Familial Hypercholesterolemia - Heterozygous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAC Score (Experimental): CAC Score evaluated by the Agatston method
  Interventions: Radiation: CAC Score

INTERVENTIONS:
Radiation: CAC Score — Computed tomography angiography (CTA) with an injection of iodine-rich contrast material

SUMMARY:
Familial hypercholesterolemia (FH) is an autosomal dominant genetic disorder characterized by elevated plasma levels of LDL-C cholesterol. This early and significant elevation of LDL-C triggers premature atherosclerosis, particularly coronary artery disease.

The initiation and management of LDL-C therapies is based on cardiovascular risk assessment. Although this is undoubtedly higher than in normocholesterolemic patients, a significant heterogeneity in heFH patients still persists that is not completely explained. Moreover, the evaluation of cardiovascular risk in patients with heFH is difficult for many reasons: non-validity of risk scores, futility of a risk calculation limited to 10 years in a young patient, late positivity of stress tests .

Therefore, there is a clear need for new cardiovascular risk assessment tools to identify higher risk heFH patients who could benefit from early and aggressive treatment.

The Coronary Artery Calcium (CAC) Score has been widely studied in the US and validated in European recommendations, and has shown the best reclassification index for patients at intermediate cardiovascular risk. A CAC score of zero is associated with a very low risk of event irrespective of the number of risk factors.

Non-calcified plaques are by definition not detected by ACC and patients with CAC = 0 may only have soft non-calcified plaques. The prevalence of these non-calcified plaques in very high-risk patients with acute coronary syndrome is 5%. The prevalence in FH patients is unknown. It has also been shown that the extent of the atherosclerotic burden is related to cardiovascular risk.

CAC score has been poorly evaluated in heFH patients. However, hypercholesterolemia and calcifications have been shown to be correlated: supra-aortic calcified masses in homozygous FH patients, early calcifications associated with chronic exposure to high LDL-C (cholesterol burden, equivalent to cigarettes) and finally, the calcifying role of statins.

The early increase of LDL-C in patients with genetic forms of FH causes premature cardiovascular damage. Investigators' hypothesis is that patients with FH have earlier coronary atheroma (and thus calcifications and non-calcified plaques) due to exposure early in life to high levels of LDL-cholesterol.

DETAILED DESCRIPTION:
The CAC score has demonstrated very powerful predictive power, particularly in asymptomatic populations.

1. The CAC score can:

   1.1- Identify subjects with high cardiovascular risk According to prospective studies, it is estimated that a CAC score> 400 is a CHD equivalent, with 10-year event rates exceeding 20% in asymptomatic patients. Prospective studies in young patients with a family history of cardiovascular disease or dyslipidaemia showed a higher risk of cardiovascular disease in those with a CAC score of 0.

   1.2- Identify subjects with low cardiovascular risk Regardless of the presence of risk factors, meta-analyses have repeatedly shown the high negative predictive power associated with a CAC = 0. The absence of calcified plaque presents an extraordinarily low risk at 10 years (1.1% at 1.7%) regardless of the number of risk factors Regardless of the presence of risk factors, meta-analyses have repeatedly shown the high negative predictive power associated with a CAC = 0 with an annual mortality rate of 0.87 compared to 1.92 in those with CAC between 1 and 10. Finally, recent studies have questioned the indication of a statin in non-HeFH patients with CAC = 0.

   Non-calcified plaques are not, by definition, detected by CAC tests and patients with CAC = 0 may only exhibit soft, non-calcified plaques. The prevalence of these non-calcified plaques in high-risk patients with acute coronary syndrome is 5% . The prevalence in heHF patients is unknown.
2. Description of the population to be studied and justification of their choice. Recruitment of patients with familial hypercholesterolemia will be carried out at the Cardiovascular Prevention Unit of the Pitié-Salpêtrière Hospital and in the Cardiology Department of Saint-Antoine Hospital. Patients will be included in the study when they come for their usual consultation or as part of their cardiovascular assessment in day hospitalization.
3. Brief description of the product (s) or experimental act (s)

   The actions and blood tests added by the research are as follows:

   Imaging: Coronary CT angiography with injection of iodinated contrast medium Biology: Calculation of cholesterol burden Vitamin D and K, estradiol, Parathormone IL-1β, IL-6, IL-11, IL-17 TGFβ1 TNFα,Genomic and proteomic analyses: Osteopontin (OPN), Osteocalcin, Osteoprotegerin, Osteonectin Receptor activator of nuclear factor kappa-B ligand, Bone morphogenetic protein 2 4 and 7, Human Bone metabolism simplicat Matrix Gla Protein MGP
4. Summary of foreseeable benefits and risks known to those who are suitable for research.

Individual risk

* Risks and physical constraints: patients will undergo a standard blood sampling for lipid levels and other biochemistry dosages and the realization of an arterial carotid and femoral ultrasound, as well as the coronary CT (with injection).
* Risks associated with the disease: there are no directly study-related risks of worsening of any previous condition in relation to the current pathology in the realization of this study. The increased cardiovascular risk associated with heFH is represented mostly by coronary artery disease which is related to the increased lifelong high cholesterol exposure.
* Risk of irradiation: study subjects wil lbe exposed to 2 - 5 mSv for the realization of both CAC score and coronary CT.
* Risk linked to the venous draining of 36 mL of blood all in all: pain, bruise, vagal faintness(malaise)
* Risks associated to the injection of iodized contrast agent: allergic reaction.

This pilot study will evaluate the prevalence of high CAC score in asymptomatic patients with heHF. This will be a first step in improving knowledge and treatment of heHF since using the CAC score, the investigators:

* Would identify the patients with increased risk to whom premature / aggressive interventions are recommended.
* Would validate a new non-invasive marker of the coronary damage in this heterogeneous population.

This project enters the wider frame of the premature ageing of the cardiovascular system with consequences on the development of cardiovascular complications such as the vascular calcifications. It was designed to highlight subclinical changes of the vascular tree to improve the treatment of the heHF and prevent the long-term complications of this disease. This project could help to identify new markers of myocardial and arterial dysfunction to propose an adapted prevention. The evaluation of the efficiency of medicine can be envisaged at the end of this study and will be encouraged by the strictly non invasive nature of the procedure as well as by its excellent reproducibility. It will also help to define strategies of prevention to improve the management of heHF.

The results will be broadcasted by means of scientific publications and of presentations in conferences or congress.

ELIGIBILITY:
Inclusion Criteria:

Patients with a heterozygous form of familial hypercholesterolemia:

* Aged 35 to 60 years old.
* Asymptomatic.
* No sign of ischemia with ECG.
* No personal history of coronary heart disease.
* Treated or untreated by cholesterol lowering treatment.
* Prior clinical examination performed
* Beneficiary of a social protection scheme or beneficiary (excluding AME)
* Informed patient and signed consent form

Exclusion Criteria:

* Person under tutorship or curatorship, or unable to give consent
* Pregnancy, breastfeeding, woman of childbearing potential in the absence of effective contraception - a urine pregnancy test will be done in hospital on the day of the coroscanner
* Contraindication to CT or injection of iodinated contrast medium or injection of esmolol hydrochloride
* Technical counter-indication: patient diameter> 70 cm, weight> 250 kg
* Renal insufficiency (CL <60)
* Personal history of cardiovascular disease and myocardial infarction
* Type 2 diabetes or uncontrolled diabetes mellitus for more than 5 years
* Uncontrolled hypertension
* Atrial fibrillation, ventricular arrhythmia
* Participation in another interventional research involving the human person or being in the exclusion period following previous research involving the human person, if applicable

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 270 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Coronary Artery Calcium evaluated by Agatston Score | one day
  Calcium Score

SECONDARY OUTCOMES:
Cholesterol burden | one day
  Total and LDL cholesterol before treatment (at diagnosis) (age at diagnosis) + yearly total and LDL-cholesterol on treatment (after diagnosis)
Coronary atheromatous plaque | one day
  Coronary computed tomography angiography: evaluation of atherosclerotic load according to the CAD-RADS classification
Peripheral atherosclerotic burden | one day
  Carotid and femoral intima-media thickness

CONTACTS AND LOCATIONS:
Overall Officials: Antonio GALLO, Dr, Principal Investigator — Hôpital Pitié-Salpêtrière, APHP
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, France